CLINICAL TRIAL: NCT04320784
Title: Effects of 4 Weeks of Time Restricted Eating Protocol on Performance, Metabolism and Blood Outcomes in Elite Cyclists
Brief Title: Effects of a Time Restricted Eating Protocol on Cyclists (TRECYC)
Acronym: TRECYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: University of Palermo (Other); University of Pavia (Other)
Responsible Party: Principal Investigator, Antonio Paoli, Full Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AP1019
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Fasting and Performance
Keywords: fasting, cyclists, athletes, time restricted eating, performance, body composition.
MeSH Terms: conditions — Fasting; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: It is a single blind, parallel arms study
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor treated anonymus data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted eating (TRE) (Experimental): TRE group consumed 100% of its estimated daily energy needs in an 8-hour time window: from 10:00 AM to 6:00 PM
  Interventions: Other: Time restricted eating
- Control (CTRL) (Active Comparator): CTRL group consumed 100% of its estimated daily energy needs in 3 meals between 7:00 AM and 9:00 PM
  Interventions: Other: Control

INTERVENTIONS:
Other: Time restricted eating — TRE group consumed 100% of its estimated daily energy needs in an 8-hour time window: from 10:00 AM to 6:00 PM
  Other Names: TRE
  Arms: Time restricted eating (TRE)
Other: Control — CTRL group consumed 100% of its estimated daily energy needs in 3 meals between 7:00 AM and 9:00 PM
  Other Names: CTRL
  Arms: Control (CTRL)

SUMMARY:
We sought to investigate the effects of 4 weeks of 16/8 time restricted eating (TRE) with windows of 16 hours of fasting and 8 hours of eating) on elite cyclists' performance, metabolic and blood parameters.

DETAILED DESCRIPTION:
Sixteen elite under-23 cyclists were randomly assigned to a TRE group or to a control group (CTRL) with a traditional meal pattern. The TRE group consumed 100% of its estimated daily energy needs in an 8-hour time window: from 10:00 AM (ante meridiem) to 6:00 PM (post meridiem) whilst the CTRL group consumed 100% of its estimated daily energy needs in 3 meals between 7:00 AM and 9:00 PM. During the experimental period, training loads were similar in the two groups. Athletes were tested before and after 4 weeks of the intervention. Body composition , basal metabolism, performances indexes and blood parameters were measured.

ELIGIBILITY:
Inclusion Criteria:

* elite under 23 cyclists male

Exclusion Criteria:

* adherence to special diets
* use of nutritional supplements (except a daily multivitamin-mineral and/or protein supplement)
* use of medications

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-06 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
VO2max | 4 weeks
  Maximal oxygen consumption (in ml O2/Kg/min) measured during a cycloergometer incremental test through a gas analyses
fat mass | 4 weeks
  fat mass measured through body impedence analyser
lean body mass | 4 weeks
  lean body mass mass measured through body impedence analyser

SECONDARY OUTCOMES:
white blood cells | 4 weeks
  white blood cells as thousands per microliter
Eosinophils | 4 weeks
  Eosinophils as percentage of total white blood cells
Monocytes | 4 weeks
  Monocytes as percentage of total white blood cells
Basophiles | 4 weeks
  Basophiles s percentage of total white blood cells
Hematocrit | 4 weeks
  Hematocrit as percentage
Haemoglobin | 4 weeks
  Haemoglobin as gram per Liter
Mean cell volume | 4 weeks
  mean cell volume as femtonLiter
mean cell haemoglobin | 4 weeks
  mean cell haemoglobin as picograms
ESR (Erythrocyte sedimentation rate ) | 4 weeks
  ESR as millimeters per hour
CRP (C-reactive protein) | 4 weeks
  CRP as milligram per deciliter
Total cholesterol | 4 weeks
  Total cholesterol as milligram per deciliter
TG (triglycerides) | 4 weeks
  TG as milligram per deciliter
glucose | 4 weeks
  glucose as milligram per deciliter
creatinine | 4 weeks
  creatinine as milligram per deciliter
creatin kinase | 4 weeks
  creatin kinase as milligram per deciliter
iron | 4 weeks
  iron as microgram per deciliter
ferritin | 4 weeks
  ferritin as microgram per liter
transferrin | 4 weeks
  ferritin as milligram per deciliter
TSH (Thyroid Stimulating Hormone) | 4 weeks
  TSH as micro international unit per milliliter
T3 (triiodothyronine) free | 4 weeks
  T3 free as picogram per milliliter
Testosterone free | 4 weeks
  Testosterone free as picogram per milliliter
IL-6 | 4 weeks
  IL-6 as picogram per milliliter
TNFalfa | 4 weeks
  TNFalfa as picogram per milliliter
IGF-1 | 4 weeks
  IGF-1 as nanogram per milliliter
Insulin | 4 weeks
  Insulin micro international unit per milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paoli A, Tinsley G, Bianco A, Moro T. The Influence of Meal Frequency and Timing on Health in Humans: The Role of Fasting. Nutrients. 2019 Mar 28;11(4):719. doi: 10.3390/nu11040719. PMID 30925707
- [Result] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674
- [Result] Tinsley GM, Forsse JS, Butler NK, Paoli A, Bane AA, La Bounty PM, Morgan GB, Grandjean PW. Time-restricted feeding in young men performing resistance training: A randomized controlled trial. Eur J Sport Sci. 2017 Mar;17(2):200-207. doi: 10.1080/17461391.2016.1223173. Epub 2016 Aug 22. PMID 27550719
- [Result] Tinsley GM, Moore ML, Graybeal AJ, Paoli A, Kim Y, Gonzales JU, Harry JR, VanDusseldorp TA, Kennedy DN, Cruz MR. Time-restricted feeding plus resistance training in active females: a randomized trial. Am J Clin Nutr. 2019 Sep 1;110(3):628-640. doi: 10.1093/ajcn/nqz126. PMID 31268131
- [Derived] Moro T, Tinsley G, Longo G, Grigoletto D, Bianco A, Ferraris C, Guglielmetti M, Veneto A, Tagliabue A, Marcolin G, Paoli A. Time-restricted eating effects on performance, immune function, and body composition in elite cyclists: a randomized controlled trial. J Int Soc Sports Nutr. 2020 Dec 11;17(1):65. doi: 10.1186/s12970-020-00396-z. PMID 33308259